CLINICAL TRIAL: NCT02346552
Title: Usability and Performance Evaluation of the AutoLap System - a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.S.T. Medical Surgery Technology LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AL-65-004
Record Dates: First submitted 2015-01-08; First posted 2015-01-27 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2016-09

CONDITIONS: General Laparoscopic Surgery Candidate; Bariatric Laparoscopic Surgery Candidate
Keywords: laparoscopic Cholecystectomy; laparoscope holder; Nissen fundoplication; paraesophageal hernia; sleeve surgery
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Procedures will be performed with the AutoLpap system used for holding and controlling the movement of the laparoscope.
  Interventions: Device: AutoLap
- Group 2 (No Intervention): Procedures will be performed with the assistance of human camera holder.

INTERVENTIONS:
Device: AutoLap
  Arms: Group 1

SUMMARY:
The main objectives of this study are to evaluate the ease of use and performance of the AutoLap system compared to human camera holder during general and bariatric laparoscopic surgeries.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Informed Consent Form (ICF).
2. Patients over 18 years who were scheduled for elective laparoscopic Cholecystectomy, Nissen fundoplication, paraesophageal hernia and sleeve surgery procedures

Exclusion Criteria:

1. Extensive adhesions that will preclude routine laparoscopic surgical approach.
2. Pregnancy
3. Patient participates in any other clinical study 60 days prior to the start of the study and throughout the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Image stability | during surgery, an expected average of 1 hour
  measured by the vibrations of inertial sensors
Usability | post surgery, an expected average of 3 minutes
  The ease of use of the AutoLap system will be evaluated by a set of questionnaires

SECONDARY OUTCOMES:
System set-up time | during surgery, an expected average of 5 minutes
Length of surgery | during surgery, an expected average of 1 hour
The Number of times that the laparoscope was removed for cleaning | during surgery, an expected average of 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Nepomnayshy, MD, Principal Investigator — Lahey Hospital & Medical Center
Locations (1):
- Lahey Hospital & Medical Center, Burlington, Massachusetts, United States